CLINICAL TRIAL: NCT06003985
Title: Assessment of Preoperative Gastric Content With Ultrasound in Patients Taking GLP1 Agonists
Brief Title: Gastric Ultrasound Assessment for Patients Taking GLP1 Agonists
Status: Completed | Type: Observational
Sponsor: Hospital for Special Surgery, New York (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-0867
Record Dates: First submitted 2023-08-15; First posted 2023-08-22 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2024-11

CONDITIONS: Gastric Ultrasound; Glucagon-like Peptide 1; Point of Care Ultrasound
Keywords: GLP1; gastric ultrasound

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control: The control group will be comprised of patients who are not currently taking any GLP-1 agonist medications. Controls will receive the ultrasound exam to assess stomach contents.
  Interventions: Other: Gastric Ultrasound Exam
- GLP-1 agonist intake: The GLP-1 agonist intake group will be comprised of patients who are currently taking any GLP-1 agonist medications. This group will receive the ultrasound exam to assess stomach contents.
  Interventions: Other: Gastric Ultrasound Exam

INTERVENTIONS:
Other: Gastric Ultrasound Exam — A gastric ultrasound is a simple, fast, non-invasive bedside diagnostic test that provides a qualitative and quantitative assessment of gastric contents. There are no known risks of a gastric ultrasound exam.

SUMMARY:
The aim of this study is to perform bedside gastric point of care ultrasound (POCUS) exams to assess the gastric volume and content (clear liquids vs solid food) perioperatively in patients who take glucagon-like peptide 1 (GLP-1) agonist medications compared to patients who do not take GLP-1 agonists.

DETAILED DESCRIPTION:
Glucagon-like peptide 1 (GLP-1) agonists have existed since 2005, however the newer once-weekly injectable medications particularly semaglutide, and tirzepatide have exploded in popularity due to their weight loss potential.

Anesthesiologists nationally have seen an increase in perioperative complications amongst patients taking these medications due to delayed gastric emptying increasing the risk of aspiration in the perioperative period. At HSS the majority of our anesthetics are done under sedation and therefore would not protect the patient from aspiration in the event of vomiting.

Protecting patients from aspiration secondary to vomiting during induction or maintenance of anesthesia has always been an important goal to make anesthesia safer leading to the development of NPO guidelines which are intended to protect against the presence of gastric content during anesthetic care. However there is growing concern that patients taking GLP-1 agonists may not be adequately protected using the current nothing by mouth or "NPO" guidelines. Up to this day there is no literature on how much gastric emptying is delayed during the use of GLP1 following the standard NPO guidelines.

Recently Gastric Ultrasound (GUS) has been introduced as a bedside tool for assessing a patients stomach contents and for the risk of aspiration. Gastric ultrasound can identify an empty stomach, a stomach filled with clear liquids, thick liquids or solid food content. If a stomach has clear liquid the volume can be calculated accurately. Generally a stomach with solid or thick liquid content or with clear liquid measuring more than 1.5 ml/kg body weight is considered a full stomach. As GUS is noninvasive and well tolerated, it offers the perfect solution to assessing patient risk in the preoperative period.

ELIGIBILITY:
Inclusion Criteria:

* GLP 1 patient group: any patient on GLP1 agonists that are dosed once per week (semaglutide, dulaglutide, tirzepatide), for all indications.
* Control group (No GLP 1 patients): any patient not on GLP1 agonists that are dosed once per week, for all indications.

Exclusion Criteria:

* patient refusal to participate
* patients with gastric bypass or any other gastric surgery
* large hiatal hernia
* patients with large ascites
* patients on peritoneal dialysis
* emergency surgery
* pre-existing diagnosis of gastroparesis

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will be comprised of patients scheduled for surgery at HSS who meet the following inclusion criteria and none of the exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 354 (Actual)
Dates: Start 2023-08-29 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-02-01 (Actual)

PRIMARY OUTCOMES:
incidence of delayed gastric emptying | This will be measured pre-operatively in the holding room area.
  delayed gastric emptying is defined by the presence of either solid food, thick liquids or a specific volume (>1.5 ml/kg) of clear liquids on gastric ultrasound.

SECONDARY OUTCOMES:
Nothing by mouth (NPO) intervals | This will be measured pre-operatively in the holding room area.
  Measure the NPO interval after last solid, liquids, and clears precisely for a subgroup analysis.
Presence of gastric peristalsis | This will be measured pre-operatively in the holding room area.
  Gastric peristalsis will be graded as present/ absent on gastric ultrasound

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Panzer, MD, Principal Investigator — Hospital for Special Surgery, Department of Anesthesiology
Locations (8):
- United States (7):
  - George Washington University Hospital, Washington D.C., District of Columbia
  - Mayo Clinic, Jacksonville, Florida
  - Albany Medical Center, Albany, New York
  - Hospital for Special Surgery, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Weill Cornell Medicine, New York, New York
  - University of Virginia, Charlottesville, Virginia
- University Health Network, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Silveira SQ, da Silva LM, de Campos Vieira Abib A, de Moura DTH, de Moura EGH, Santos LB, Ho AM, Nersessian RSF, Lima FLM, Silva MV, Mizubuti GB. Relationship between perioperative semaglutide use and residual gastric content: A retrospective analysis of patients undergoing elective upper endoscopy. J Clin Anesth. 2023 Aug;87:111091. doi: 10.1016/j.jclinane.2023.111091. Epub 2023 Mar 2. PMID 36870274
- [Background] Maselli DB, Camilleri M. Effects of GLP-1 and Its Analogs on Gastric Physiology in Diabetes Mellitus and Obesity. Adv Exp Med Biol. 2021;1307:171-192. doi: 10.1007/5584_2020_496. PMID 32077010
- [Background] Nakatani Y, Maeda M, Matsumura M, Shimizu R, Banba N, Aso Y, Yasu T, Harasawa H. Effect of GLP-1 receptor agonist on gastrointestinal tract motility and residue rates as evaluated by capsule endoscopy. Diabetes Metab. 2017 Oct;43(5):430-437. doi: 10.1016/j.diabet.2017.05.009. Epub 2017 Jun 23. PMID 28648835